CLINICAL TRIAL: NCT00736151
Title: A Phase II, Multicentre, Pilot, Randomised, Double Blind Placebo Controlled Dose Titration Study to Evaluate the Safety, Maximum Tolerated Dose and Preliminary Evidence of Efficacy of Orally Administered Ralfinamide at Four Doses (80, 160, 240 and 320 mg/Day) in Patients With Neuropathic Pain
Brief Title: Phase II Dose Titration Study in Patients With Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Stefano Rossetti, MD, Newron Pharmaceuticals S.p.A
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NW-1029/001/II/2003; EUDRACT Number 2004-000557-35
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Ralfinamide

ARMS (2):
- 1 (Experimental): Ralfinamide administered orally at rising doses of 80 - 320 mg/day
  Interventions: Drug: Ralfinamide
- 2 (Active Comparator): Placebo controlled with randomization of 2:1
  Interventions: Drug: Ralfinamide

INTERVENTIONS:
Drug: Ralfinamide — Oral tablets administered at rising doses of 80 - 320 mg/day

SUMMARY:
The purpose of this study is to examine the effects of various increasing doses of Ralfinamide in patients with neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Females post-menopausal for at least 12 months, 24 months in India, Poland, and Austria
* Diagnosed by neurologist with current neuropathic pain

Exclusion Criteria:

* See inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2004-05; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change of pain intensity | Baseline to week 8 or last visit

SECONDARY OUTCOMES:
The incidence of adverse events | From baseline to week 8 or last visit

CONTACTS AND LOCATIONS:
Locations (47):
- Austria (4):
  - Universitatsklinik Fur Neurologie, Graz
  - Universitatsklinik Fur Neurologie, Innsbruck
  - LKH, Klagenfurt
  - General Hospital AKH, Vienna
- Czechia (6):
  - Fakultni nemocnice u svate' Anny v Brne, Brno
  - Fakultni nemocnice Brno, Brno-Bhunice
  - University Hospital Olomouc, Olomouc
  - Univercity Hospital Pilsen, Pizen
  - Fakultni Thomayerova nemocnices poliklinikou, Prague
  - Na Homolce Hospital, Prague
- India (10):
  - Neurology Centre, Ahmedabad
  - M.S. Ramaiah Medical, Bangalore
  - R.S. R'S Trinity Acute Care Hospital, Chennai
  - Sri Ramachandra medical College, Chennai
  - Care Hospital, Hyderabad
  - Chowpatty Medical Centre, Mumbai
  - Brain and Mind Institute, Nagpur
  - Apollo Hospital, Pradesh
  - Brain Waves Clinic, Pune
  - Vijaya Health Centre, Vadapalani
- Italy (15):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ce. S.I. Fondazione Universitaria, Chieti
  - Ospedale Clinicizzato Universitario SS. Annunziata, Chieti
  - Arcispedale Sant'Anna, Ferrara
  - Azienda Ospedaliera San Martino, Genova
  - Universita degli Studi di Genova, Genova
  - Ospedale Luigi Sacco, Grassi
  - Ospedale Civile Umberto I, Mestre
  - Ospedale San Raffaele, Milan
  - Istituto Scientifico di Riabilazione di Montescano, Montescano
  - Policlinico Universitario Federico II, Napoli
  - UCADH, Pavia
  - Presidio Ospedaliero Monteluce, Perugia
  - Universita degli Studi di Roma, Roma
  - Policlinico G.B. Rossi, Verona
- Poland (8):
  - Centrum Medyczne Osteomed, Bialobrzeska
  - Centrum Kliniczno Badawcze, Elblag
  - Wojewodzki Szpiyal Spejalistyczny, Gdansk
  - Center Of Clinical Neurology, Krakow
  - Osrodek Baden Klinicznych, Lublin
  - Wojskowy Instytut Medyczny, Warsaw
  - Wroclaw Medical University, Wroclaw
  - Oddzial Neurologiczny, Zgierz
- United Kingdom (4):
  - Gartnavel General Hospital, Glasgow
  - Barta and The London NHS Trust, London
  - Kings College Hospital, London
  - Solihull Hospital, West Midlands